CLINICAL TRIAL: NCT05694234
Title: Influences of Sugammadex on Postoperative Progress in Patients With Myasthenia Gravis Undergoing Video-assisted Thoracoscopic Thymectomy: Retrospective Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2021-0560
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sugammadex group: patients who administered sugammadex
- AChEI group: patients who administered pyridostigmine-glycopyrrolate or neostigmine-glycopyrrolate

SUMMARY:
"Several case reports have described the use of rocuronium and sugammadex in patients with myasthenia gravis (MG). However, reports regarding the effects of sugammadex compared with that of acetylcholinesterase inhibitors (AChEIs) on perioperative outcomes of video-assisted thoracoscopic surgery (VATS)-thymectomy in patients with MG are still lacking. Thus, the investigators will investigate the effects of sugammadex compared to AChEIs on the postoperative recovery in patients with MG who underwent VATS-thymectomy.

This retrospective study include patients with MG, aged> 18 years who received sugammadex or pyridostigmine-glycopyrrolate or neostigmine-glycopyrrolate after VATS-thymectomy between November 2007 and December 2020. Inverse Probability of Treatment Weighting (IPTW) adjustment will be performed to balance the baseline characteristics between the two groups. The primary outcome is the length of postoperative hospital stay, and the secondary outcomes are the incidence of postoperative mortality and postoperative complications, as well as postoperative extubation and reintubation rates in the operating room after VATS-thymectomy; the outcomes are compared between the two groups. "

ELIGIBILITY:
Inclusion Criteria:

* patients underwent VATS-thymectomy between November 2007 and December 2020

Exclusion Criteria:

* Patients who was not diagnosed with myasthenia gravis
* Age ≤ 18
* Patients for which no reversal agent was used

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myasthenia gravis who underwent video-assisted thoracoscopic thymectomy
Sampling Method: Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
hospital stay | up to 1 year
  length of postoperative hospital stay (day)

SECONDARY OUTCOMES:
incidence of postoperative mortality | up to 1 year
postoperative complication incidence | up to 1 year
postoperative extubation rate in the OR | up to 1 year
postoperative reintubation rate in the OR | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Na Young Kim, Principal Investigator — Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 3years